CLINICAL TRIAL: NCT06923098
Title: PET/CT GUIDED BIOPSY VERSUS CT GUIDED BIOPSY IN EVALUATION OF SUSPECTED LUNG NEOPLASMS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: All India Institute of Medical Sciences, Bhubaneswar (Other)
Responsible Party: Principal Investigator, Girish Kumar Parida, Assistant Professor, All India Institute of Medical Sciences, Bhubaneswar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IEC/AIIMS BBSR/PG Thesis/2023-
Record Dates: First submitted 2025-04-04; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Lung Diseases
Keywords: CT guided biopsy; PET-CT guided biopsy; Lung lesions
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CT guided biopsy (Active Comparator)
  Interventions: Procedure: CT guided biopsy
- PET-CT guided biopsy (Experimental)
  Interventions: Procedure: PET-CT guided biopsy

INTERVENTIONS:
Procedure: PET-CT guided biopsy — PET-CT guided biopsy of lung lesions
  Arms: PET-CT guided biopsy
Procedure: CT guided biopsy — CT guided biopsy of lung lesions
  Arms: CT guided biopsy

SUMMARY:
Percutaneous CT guided biopsy is a well-established, standard sampling technique for suspected neoplastic lesions located in peripheral region in lung parenchyma. Inconclusive results on CT guided biopsy is substantially higher in large lung lesions which are prone to cause peripheral pneumonia, atelectasis and even regional necrosis, which are hard to be distinguished from tumor on CT images.

Functional imaging guided biopsy like PET/CT guided biopsy identifies areas of highest concentration of neoplastic cells and provides accurate results. Only a few studies have been done regarding PET/CT guided biopsy and studies omparing PET/CT guided and CT guided percutaneous transthoracic lung biopsy are very few and this study would be a randomized trial comparing these diagnostic modalities in terms of diagnostic yield, diagnostic accuracy of sample and complications.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years
* INR < 1.2 and platelet counts > 80,000/mm3
* CT thorax with lung lesion more than 10 mm.
* Accessible lesions for CT-guided biopsy.

Exclusion Criteria:

* Participants with pre-existing bleeding diathesis like hemophilia, coagulopathy defined by -INR ≥1.2 and Platelet counts ≤ 80,000/mm3
* Participants who refuse to provide consent
* Signs of hypoperfusion like hypotension, cyanosis etc.
* Presence of hypoxemia with SpO2 < 94 %- measured in a pulse oximeter)
* Pregnant/Lactating female subjects
* Non-cooperative subjects
* Lesions that are inaccessible (decision made on pre-biopsy planning)
* Serum creatinine level more than 2mg/dl.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Inconclusive pathology findings | 1 month
  Comparing the proportion of inconclusive pathology reports in both arms

SECONDARY OUTCOMES:
Incidence of pneumothorax and hemoptysis | 1 month
  Incidence of pneumothorax and hemoptysis in both arms

CONTACTS AND LOCATIONS:
Locations (1):
- All India Institute of Medical Sciences, Bhubaneswar, Bhubaneswar, Odisha, India